CLINICAL TRIAL: NCT01784757
Title: A Bioavailability Study of ODM-201 Formulations With a Safety and Tolerability Extension Component in Subjects With Metastatic Chemotherapy-naive Castration-resistant Prostate Cancer
Brief Title: Bioavailability Study of ODM-201 in Subjects With Metastatic Chemotherapy-naive Castration-resistant Prostate Cancer
Acronym: ARAFOR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 3104003; 2012-002279-32 (EudraCT Number)
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ODM-201 Tablet A (Experimental): ODM-201 tablet A in fed and fasted states plus ODM-201 capsule in fed state in randomised order.
  Interventions: Drug: ODM-201 Tablet A; Drug: ODM-201 capsule formulation
- ODM-201 Tablet B (Experimental): ODM-201 Tablet B in fed and fasted states plus ODM-201 capsule in fed state in randomised order.
  Interventions: Drug: ODM-201 Tablet B; Drug: ODM-201 capsule formulation

INTERVENTIONS:
Drug: ODM-201 Tablet A — Tablet A formulation of ODM-201
  Arms: ODM-201 Tablet A
Drug: ODM-201 Tablet B — Tablet B formulation of ODM-201
  Arms: ODM-201 Tablet B
Drug: ODM-201 capsule formulation — Capsule formulation of ODM-201

SUMMARY:
A study to investigate which of two different tablet formulations of ODM-201 is best suited for use in the further development of the compound in the treatment of metastatic chemotherapy-naive castration-resistant prostate cancer. Patients successfully completing the bioavailability study will be able to receive further treatment with the current capsule formulation of ODM-201 until progression of their disease with the safety and tolerability of ODM-201 being assessed throughout.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained.
* Histologically confirmed adenocarcinoma of prostate
* Progressive metastatic disease
* Ongoing androgen deprivation therapy with a luteinising hormone-releasing hormone (LHRH) analogue or antagonist or bilateral orchiectomy
* Adequate bone marrow, hepatic and renal function
* Able to swallow the ODM-201 whole as a capsule or tablet.

Exclusion Criteria:

* Previous chemotherapy for prostate cancer.
* Known metastases in the brain.
* History of other malignancy within the previous 5 years, except a basal cell carcinoma of skin.
* Known gastrointestinal condition that can significantly affect the absorption of the study treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of ODM-201 | 0-48 hrs
  The area under the concentration-time curve from time zero to the last sample with the quantifiable concentration calculated with linear trapezoidal rule.
Cmax of ODM-201 | 0-48 hrs
  The plasma peak concentration.

SECONDARY OUTCOMES:
tmax of ODM-201 | 0-48 hrs
  The time to reach peak concentration.
Terminal elimination rate constant of ODM-201 | 0-48 hrs
  The terminal elimination rate constant from log-linear portion of a concentration-time curve.
Terminal elimination half-life of ODM-201 | 0-48 hrs
  The terminal elimination half-life that will be calculated with the equation ln2/terminal elimination rate constant.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Fizazi, MD PhD, Principal Investigator — Institut Gustave Roussy, University of Paris
Locations (1):
- P. Stradina Clinical University Hospital, Riga, Latvia

REFERENCES:
- [Derived] Shore ND, Tammela TL, Massard C, Bono P, Aspegren J, Mustonen M, Fizazi K. Safety and Antitumour Activity of ODM-201 (BAY-1841788) in Chemotherapy-naive and CYP17 Inhibitor-naive Patients: Follow-up from the ARADES and ARAFOR Trials. Eur Urol Focus. 2018 Jul;4(4):547-553. doi: 10.1016/j.euf.2017.01.015. Epub 2017 Feb 14. PMID 28753851